CLINICAL TRIAL: NCT05458063
Title: The Effectiveness of the Urine Mitochondrial Deoxyribonucleic Acid and, Serum Beta 2 Microglobulin as a Biomarker of Renal Function Impairment in Critically Ill Surgical Patients
Brief Title: The Effectiveness of Urine mtDNA and Beta 2-MG to Predict Acute Kidney Injury for Critically Ill Surgical Patients
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Kwangmin Kim, Clinical assistant professor, Wonju Severance Christian Hospital
Other Study IDs: BMPAS2022; 2022R1I1A1A01069511 (Other Grant/Funding Number: National Research Foundation of Korea)
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Surgery-Complications; Acute Kidney Injury; Critical Illness
Keywords: Critically ill surgical patient; Acute kidney injury; Urine mitochondrial DNA; Beta 2-microglobulin; Biomarker
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell free mitochondrial DNA in urine is released from renal parenchymal cells, and tubular cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted in Surgical intensive care unit and trauma intensive care unit: all surgical patients who planned to admit in surgical and trauma intensive care unit in emergency room

SUMMARY:
1. Research background

1. Research hypothesis The development of acute kidney injury (AKI) can be predicted using urine mitochondrial deoxyribonucleic acid (UmtDNA), serum and urine beta-2 microglobulin (β2-MG) in critically ill surgical patients
2. Basis of research hypothesis

   i. Correlation between mitochondria and renal function (Results of previous studies)
   * Mitochondria are involved in development and recovery of diabetic nephropathy.
   * UmtDNA can be used as early marker to detect the development of AKI

     ※ Mitochondria
   * As an organelle located within the cell, it is an organ that produces energy through adenosine triphosphate (ATP) through cellular oxidative phosphorylation.
   * The kidney has the second most mitochondria after the heart.

   II. Correlation between elevation of β2-MG and renal function
   * Circulating β2-MG infiltrates the glomerulus and is reabsorbed and metabolized in the proximal tubule of the kidney. Therefore, it increases in the blood due to a decrease in metabolism when renal function is abnormal.

     ※ Beta 2-microglobulin
   * As the light chain of the class I major histocompatibility antigen, it is a protein distributed in nucleated cells (especially lymphocytes and monocytes) in the body.

   III. Mechanism of acute kidney injury in critically ill surgical patients
   * Blood flow to the kidneys is reduced due to decreased cardiac output, vasoconstriction due to systemic inflammatory response, hemodynamic changes, and decreased body fluid. This leads to renal tubular injury along with ischemic reperfusion injury.
   * Renal tubular injury increases the permeability of the transition pore that connects the outer and inner mitochondrial membranes, resulting in mitochondrial structural damage and oxidative injury. It causes a decrease of ATP in kidney cells and induces apoptosis of kidney cells.
   * Urine mtDNA, a product of this kidney injury, could be used as a biomarker to predict impairment of renal function in critically ill surgical patients.
   * Serum β2-MG maybe increase due to a decrease of metabolism of β2-MG in AKI.

DETAILED DESCRIPTION:
1. Research objective

1. Demonstrate of the association between urine mitochondrial deoxyribonucleic acid copy number (UmtDNAcn), beta 2-microglobulin (β2-MG) and acute kidney injury in critically ill surgical patients
2. Demonstrate of the effectiveness of UmtDNAcn and β2-MG as a biomarker to predict AKI development and recovery

2. Contents of the research project.

1. Analysis of correlation between UmtDNAcn, β2-MG and development of AKI

   * Verifying the correlation between UmtDNAcn and blood β2-MG measured at the initial presentation and patients diagnosed AKI according to the Acute Kidney Injury Network (AKIN) criteria.
2. Analysis of correlation between UmtDNAcn, β2-MG and recovery of AKI

   * Verifying the correlation between UmtDNAcn and blood β2-MG measured at the initial presentation and AKI recovery
   * AKI recovery was defined as the case when the AKI stage according to the AKIN criteria on the 7th day of AKI onset was reduced from AKI stage measured at the beginning of the AKI onset.
3. Comparison with other biomarkers (delta neutrophil index, creatinine, cystatin C) - Comparison of sensitivity and specificity of UmtDNAcn, β2-MG, and other biomarkers previously used such as creatinine, cystatin C, and delta neutrophil index.

3. Strategies and methods for the research project

1. subject: all surgical patients who planned to admit surgical and trauma intensive care unit in emergency room
2. Study period and patient recruitment i. 1st and 2nd year

   * 120 patients
3. Measurement of UmtDNAcn, β2-MG i. urine and blood sampling: at the initial presentation and again on hospital say #1 and #3
4. Analysis of correlation between UmtDNAcn, β2-MG and AKI development, recovery

   i. Statistical analysis of UmtDNAcn, β2-MG measured at the initial presentation, on hospital day #1, and #3 between patients with no AKI and AKI

   ii. Statistical analysis of UmtDNAcn, β2-MG measured at the initial presentation, on hospital day #1, and #3 between patients with no AKI recovery and AKI recovery

   ※ AKI recovery was defined as the case when the AKI stage according to the AKIN criteria on the 7th day of AKI onset was reduced from AKI stage measured at the beginning of the AKI onset.

   iii. Comparison with other biomarkers (delta neutrophil index, creatinine, cystatin C)
   * Comparison of sensitivity and specificity to predict AKI of UmtDNAcn, β2-MG, and other biomarkers previously used such as creatinine, cystatin C, and delta neutrophil index measure at the initial presentation, on hospital day #1 and #3. .

ELIGIBILITY:
Inclusion Criteria:

* All surgical patients who planned to admit to surgical and trauma intensive care unit in emergency room

Exclusion Criteria:

* Age ≤18 years
* Pregnancy in women
* Chronic kidney disease history
* Death at initial presentation of the case

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All surgical patients who planned to admit to surgical and trauma intensive care unit in emergency room
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury (dichotomous) | Within 30 days after ICU admission
  Acute kidney injury according to Acute Kidney Injury Network (AKIN) criteria
Acute kidney injury recovery (dichotomous) | Within 30 days after ICU admission
  the case when the AKI stage according to the AKIN criteria on the 7th day of AKI onset was reduced from AKI stage measured at the beginning of the AKI onset

SECONDARY OUTCOMES:
Mortality (dichotomous) | Within 30 days after ICU admission
  The number of deaths
Hospital length of stay (continuous) | From date of the admission until the date of first discharge from the hospital, assessed up to 60 days
  Measured in days from admission to discharge
Intensive care unit (ICU) stay (continuous) | From date of ICU admission (in cases of ICU admission at the initial presentation) until the date of first discharge from ICU, assessed up to 60 days
  Measured in days from ICU admission to ICU out

CONTACTS AND LOCATIONS:
Overall Officials: In Sik Shin, Principal Investigator — Wonju Severance Christian Hospital
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pagliarini DJ, Calvo SE, Chang B, Sheth SA, Vafai SB, Ong SE, Walford GA, Sugiana C, Boneh A, Chen WK, Hill DE, Vidal M, Evans JG, Thorburn DR, Carr SA, Mootha VK. A mitochondrial protein compendium elucidates complex I disease biology. Cell. 2008 Jul 11;134(1):112-23. doi: 10.1016/j.cell.2008.06.016. PMID 18614015
- [Background] Chang CC, Chiu PF, Wu CL, Kuo CL, Huang CS, Liu CS, Huang CH. Urinary cell-free mitochondrial and nuclear deoxyribonucleic acid correlates with the prognosis of chronic kidney diseases. BMC Nephrol. 2019 Oct 28;20(1):391. doi: 10.1186/s12882-019-1549-x. PMID 31660901
- [Background] Cha SW, Shin IS, Kim DG, Kim SH, Lee JY, Kim JS, Yang JW, Han BG, Choi SO. Effectiveness of serum beta-2 microglobulin as a tool for evaluating donor kidney status for transplantation. Sci Rep. 2020 May 15;10(1):8109. doi: 10.1038/s41598-020-65134-6. PMID 32415140
- [Background] Whitaker RM, Stallons LJ, Kneff JE, Alge JL, Harmon JL, Rahn JJ, Arthur JM, Beeson CC, Chan SL, Schnellmann RG. Urinary mitochondrial DNA is a biomarker of mitochondrial disruption and renal dysfunction in acute kidney injury. Kidney Int. 2015 Dec;88(6):1336-1344. doi: 10.1038/ki.2015.240. Epub 2015 Aug 19. PMID 26287315
- [Background] Hu Q, Ren J, Ren H, Wu J, Wu X, Liu S, Wang G, Gu G, Guo K, Li J. Urinary Mitochondrial DNA Identifies Renal Dysfunction and Mitochondrial Damage in Sepsis-Induced Acute Kidney Injury. Oxid Med Cell Longev. 2018 Feb 26;2018:8074936. doi: 10.1155/2018/8074936. eCollection 2018. PMID 29682165
- [Background] Trongtrakul K, Sawawiboon C, Wang AY, Chitsomkasem A, Limphunudom P, Kurathong S, Prommool S, Trakarnvanich T, Srisawat N. Acute kidney injury in critically ill surgical patients: Epidemiology, risk factors and outcomes. Nephrology (Carlton). 2019 Jan;24(1):39-46. doi: 10.1111/nep.13192. PMID 29124867